CLINICAL TRIAL: NCT01497444
Title: Study of Sorafenib + TH-302: Phase I in Advanced Renal Cell Carcinoma (RCC) and Advanced Hepatocellular Carcinoma (HCC) and Phase II in 1st Line Advanced HCC
Brief Title: Sorafenib Tosylate and Hypoxia-Activated Prodrug TH-302 in Treating Patients With Advanced Kidney Cancer or Liver Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N1153; NCCTG-N1153; CDR0000720022 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-00095 (Registry Identifier: CTRP (Clinical Trials Reporting System)); U10CA031946 (NIH)
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Kidney Cancer; Liver Cancer
Keywords: recurrent adult primary liver cancer; recurrent renal cell cancer; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Renal Cell | interventions — TH 302; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib and TH-302 (Experimental): Patients will be administered sorafenib tablets to take twice daily by mouth, every day of each cycle. Patients will also be given TH-302 intravenously (IV) on days 8, 15 and 22 of each cycle. A cycle is 28 days.
  Interventions: Drug: hypoxia-activated prodrug TH-302; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: hypoxia-activated prodrug TH-302
Drug: sorafenib tosylate

SUMMARY:
RATIONALE: Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth by blocking blood flow to the tumor. Drugs used in chemotherapy, such as hypoxia-activated prodrug TH-302, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib tosylate together with hypoxia-activated prodrug TH-302 may kill more tumor cells.

PURPOSE: This phase I/II trial studies the side effects and best dose of giving sorafenib tosylate together with hypoxia-activated prodrug TH-302 and to see how well they work in treating patients with advanced kidney cancer or liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose (MTD) and recommended Phase II dosing (RP2D) for the combination of sorafenib tosylate and hypoxia-activated prodrug TH-302 (TH-302) in patients with hepatocellular carcinoma (HCC) and renal cell carcinoma (RCC; non-HCC) advanced solid tumors. (Phase I)
* To evaluate the overall response rate (RR) determined based on modified RECIST criteria (Lencioni and Llovet 2010) in patients with advanced HCC receiving sorafenib tosylate with TH-302. (Phase II)

Secondary

* To characterize overall toxicity profile of sorafenib tosylate + TH-302 within patients with HCC and RCC (non-HCC) advanced solid tumors. (Phase I)
* To characterize the responses of sorafenib tosylate + TH-302 within patients with HCC and RCC (non-HCC) advanced solid tumors. (Phase I)
* To assess the adverse events (AEs) profile and safety profile of sorafenib tosylate in combination with TH-302 in patients with advanced HCC. (Phase II)
* To estimate the overall response rate based on standard RECIST criteria in the study population. (Phase II)
* To estimate the duration of response based on modified (standard) RECIST criteria in the study population. (Phase II)
* To estimate the progression free survival (PFS) in the study population. (Phase II)
* To estimate the overall survival (OS) in the study population. (Phase II)
* To estimate the alpha-fetoprotein (AFP) response rate (defined as > 20% decrease of AFP from baseline) in the study population. (Phase II)

OUTLINE: This is a multicenter, phase I dose-escalation study followed by a phase II study.

Patients receive sorafenib tosylate orally (PO) twice daily (BID) on days 1-28 and hypoxia-activated prodrug TH-302 IV over 30 minutes on days 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Some patients undergo blood sample collection periodically during study for alpha-fetoprotein analysis.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Phase I Registration - Inclusion Criteria

* Age ≥18 years
* Cytological or histological confirmed diagnosis of advanced hepatocellular or renal cell carcinoma. HCC patients should not be amenable to treatment with surgery or to orthotopic liver transplant.
* Patients must have measurable disease as defined in the protocol.
* RCC patients only: Tumor progression after receiving standard/approved chemotherapy and/or targeted agent, where there is no approved therapy or for tumors where sorafenib based therapy would be standard therapy.
* HCC patients only:

  * First line (i.e., no prior systemic therapy) or second line (with prior first line sorafenib therapy only) advanced HCC.
  * Child Pugh class A or B7 liver disease
  * Prior chemoembolization, radioembolization, radiofrequency ablation (RFA), or other local ablative therapies are permissible if ≥6 weeks from procedure with evidence of progression or new metastatic disease, if applicable.
* ECOG Performance Status (PS) 0 or 1.
* The following laboratory values obtained ≤14 days prior to registration.

  * Absolute neutrophil count (ANC) ≥1200/mm3
  * Peripheral Platelet Count (PLT) ≥75,000/mm3
  * Hemoglobin (HgB) >8.5 g/dL
  * Bilirubin ≤3.0 x upper limit of normal (ULN)
  * SGOT (AST) ≤2.5 x ULN, if subject has HCC or liver metastases ≤5 x UL
  * SGPT (ALT) ≤2.5 x ULN, if subject has HCC or liver metastases ≤5 x ULN
  * Creatinine ≤1.5 x ULN
  * INR ≤1.5 x ULN. Patients receiving anti-coagulation therapy are permitted as long as they have a stable INR≤3.0.
* Negative pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.

  * Provide informed written consent.
  * Willing to return to Alliance enrolling institution for follow-up.
  * Life expectancy ≥3 months.

Phase I Registration - Exclusion Criteria

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown.

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception for the duration of study participation. Men and women should continue to use adequate birth control after the last administration of sorafenib and TH-302 under the guidance of their treating physician.
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Receiving any other investigational agent.
* Other active malignancy ≤3 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix. NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer.
* Inadequately controlled hypertension (systolic blood pressure of >150 mmHg or diastolic pressure >100 mmHg on anti-hypertensive medications).
* Major surgical procedures, or significant traumatic injury ≤14 days prior to registration or anticipation of need for elective or planned major surgical procedure during the course of the study.
* New York Heart Association (NYHA) classification III or IV congestive heart failure.
* Received treatment with radiation therapy or investigational therapy ≤28 days prior to registration.
* RCC patients only: Having received chemotherapy prior to study entry within 5 half-lives of the agent (as described in the package insert), or 4 weeks prior to registration (whichever is shorter) with resolution of side effects from therapy to ≤grade 1.
* Known central nervous system or brain metastasis that are either symptomatic or untreated. Note: Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.

  * Note: Subjects with CNS metastases that have been treated and are stable without symptoms for ≥ 4 weeks after completion of treatment are eligible.
* HCC patients only: Cancer potentially amenable to local modalities of therapy or surgical resection.
* Known or suspected allergy or hypersensitivity to any component of TH-302, sorafenib, or any of the sorafenib excipients.
* Any condition that severely impairs patient's ability to swallow whole pills.
* QTc interval >500 msec on baseline EKG.
* Documented history of prolonged QTc interval ≤ 6 months prior to registration.
* Receiving any medication that has documented data or is generally accepted as having increased risk of QT prolongation and/or Torsades de Pointes.
* Receiving any medications or substances that are inducers or strong or moderate inhibitors of CYP3A4, see the protocol for a complete listing.
* Fibrolamellar histology HCC, mixed hepatocholangiocarcinoma, hepatic sarcomas and other non-HCC primary liver tumors.
* History of lobectomy involving >50% of lobe.
* Radioembolization within 8 weeks of Day 1 dosing of sorafenib.

Phase II Registration - Inclusion Criteria

* Age ≥18 years
* Cytological or histological confirmed diagnosis of hepatocellular carcinoma that is locally advanced or metastatic and is not amenable to treatment with surgery or to orthotopic liver transplant.
* Patients must have measurable disease as defined in Section 11.0 must have at least one non-nodal lesion.
* First line advanced HCC (i.e., no prior systemic therapy).
* Child Pugh class A or B7 liver disease
* Prior chemoembolization, radioembolization, radiofrequency ablation (RFA), or other local ablative therapies are permissible if ≥6 weeks from procedure with evidence of progression or new metastatic disease, if applicable.
* ECOG Performance Status (PS) 0 or 1.
* The following laboratory values obtained ≤14 days prior to registration.

  * Absolute neutrophil count (ANC) ≥1200/mm^3
  * Peripheral Platelet Count (PLT) ≥75,000/mm^3
  * Hemoglobin (HgB) >8.5 g/dL
  * Total bilirubin ≤3.0 x upper limit of normal (ULN)
  * SGOT (AST) ≤5 x ULN.
  * SGPT (ALT) ≤5 x ULN.
  * Creatinine ≤1.5 x ULN.
  * INR ≤1.5 x ULN. Patients receiving anti-coagulation therapy are permitted as long as they have a stable INR≤3.0.
* Negative pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.
* Provide informed written consent.
* Willing to return to Alliance enrolling institution for follow-up.
* Life expectancy ≥3 months.
* Ability to receive intravenous contrast for the purpose of imaging.

Phase II Registration - Exclusion Criteria

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown.

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception for the duration of study participation. Men and women should continue to use adequate birth control after the last administration of sorafenib and TH-302 under the guidance of their treating physician.
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Receiving any other investigational agent.
* Other active malignancy ≤3 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix. NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer.
* Inadequately controlled hypertension (systolic blood pressure of >150 mmHg or diastolic pressure >100 mmHg on anti-hypertensive medications).
* Major surgical procedures, or significant traumatic injury ≤14 days prior to registration or anticipation of need for elective or planned major surgical procedure during the course of the study.
* New York Heart Association (NYHA) classification III or IV congestive heart failure.
* Received treatment with radiation therapy or investigational therapy ≤28 days prior to registration.
* Known central nervous system or brain metastasis that are either symptomatic or untreated. Note: Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.

  * Note: Subjects with CNS metastases that have been treated and are stable without symptoms for ≥ 4 weeks after completion of treatment are eligible.
* Fibrolamellar histology HCC, mixed hepatocholangiocarcinoma, hepatic sarcomas and other non-HCC primary liver tumors.
* Cancer potentially amenable to local modalities of therapy or surgical resection.
* Known or suspected allergy or hypersensitivity to any component of TH-302, sorafenib, or any of the sorafenib excipients
* Any condition that severely impairs patient's ability to swallow whole pills.
* QTc interval >500 msec on baseline EKG.
* Documented history of prolonged QTc interval ≤ 6 months prior to registration.
* Receiving any medication that has documented data or is generally accepted as having increased risk of QT prolongation and/or Torsades de Pointes.
* Receiving any medications or substances that are inducers or strong or moderate inhibitors of CYP3A4, please see protocol for a complete listing.
* History of lobectomy involving >50% of lobe.
* Radioembolization within 8 weeks of Day 1 dosing of sorafenib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Number of dose-limiting toxicity incidents as assessed by CTCAE version 4.0 (Phase I) | Up to 24 weeks
MTD of sorafenib tosylate and TH-302 (Phase I) | Up to 24 weeks
Overall response rate (Phase II) | Up to 3 years

SECONDARY OUTCOMES:
Adverse events as assessed by NCI CTCAE version 4.0 (Phase II) | Up to 3 years
Overall response rate based on standard RECIST criteria (Phase II) | Up to 3 years
Duration of response based on modified (standard) RECIST criteria (Phase II) | Up to 3 years
PFS (Phase II) | Up to 3 years
OS (Phase II) | Up to 3 years
AFP response rate (Phase II) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh J. Borad, MD, Study Chair — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic Cancer Center, Rochester, Minnesota